CLINICAL TRIAL: NCT05814835
Title: First in Human Study of 68Ga/64Cu-FAPI-XT117 PET/CT in Patients With Malignant
Brief Title: First in Human Study of 68Ga/64Cu-FAPI-XT117 PET/CT in Patients With Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Principal Investigator, Ruimin Wang, chief of nuclear medicine department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XT-XTR016-1-01
Record Dates: First submitted 2023-03-03; First posted 2023-04-18 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Malignant Solid Tumors
Keywords: 68Ga-FAPI 64Cu-FAPI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga/64Cu-FAPI-XT117 PET/CT (Experimental): Each patient will receive 2-4 mCi, 4-6 mCi or 6-8 mCi 68Ga/64Cu-FAPI-XT117 intravenously (IV), and then PET/CT scanning within the specified time. On another day, patients receive 18F-FDG and then undergo PET/ CT.
  Interventions: Drug: 2-4 mCi 68Ga/64Cu-FAPI-XT117; Drug: 4-6 mCi 68Ga/64Cu-FAPI-XT117; Drug: 6-8 mCi 68Ga/64Cu-FAPI-XT117

INTERVENTIONS:
Drug: 2-4 mCi 68Ga/64Cu-FAPI-XT117 — 68Ga/64Cu-FAPI-XT117 and 18F-FDG PET/CT were performed for each patient(the interval was more than one day and less than four weeks). PET/CT images were acquired 30min, 60min, 120min after 2-4 mCi 68Ga/64Cu-FAPI-XT117 injection.
Drug: 4-6 mCi 68Ga/64Cu-FAPI-XT117 — 68Ga/64Cu-FAPI-XT117 and 18F-FDG PET/CT were performed for each patient(the interval was more than one day and less than four weeks). PET/CT images were acquired 30min, 60min, 120min after 4-6 mCi 68Ga/64Cu-FAPI-XT117 injection.
Drug: 6-8 mCi 68Ga/64Cu-FAPI-XT117 — 68Ga/64Cu-FAPI-XT117 and 18F-FDG PET/CT were performed for each patient(the interval was more than one day and less than four weeks). PET/CT images were acquired 30min, 60min, 120min after 6-8 mCi 68Ga/64Cu-FAPI-XT117 injection.

SUMMARY:
This is the first-in-human study of 68Ga/64Cu-FAPI-XT117, which is an prospective, single-arm phase I clinical study.

DETAILED DESCRIPTION:
20 patients with confirmed diagnosis of malignant solid tumor by histopathology or clinical judgment and required routine 18F-FDG PET/CT imaging were recruited. 68Ga/64Cu-FAPI-XT117 and 18F-FDG PET/CT were performed for each patient in any order(the interval was more than one day and less than four weeks). They were assigned to three 68Ga/64Cu-FAPI-XT117 dose groups, including 3±10% mCi、5±10% mCi and 7 ±10% mCi. PET/CT images were acquired 30min, 60min, 120min after injection. The primary end point was safety, secondary endpoints were accuracy (AC), sensitivity (SE), specificity (SP), positive predictive value (PPV), and change in management. Exploring end point was image quality, including qualitative and quantitative evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 1. signed the informed consent
* 2. ≥18 years old
* 3. confirmed as malignant solid tumor by histopathology or clinical judgment
* 4. Patients will undergo 18F-FDG PET/CT examination

Exclusion Criteria:

* 1. Known allergy to components of the investigational drug or its analogues
* 2. suspected to have a certain disease or condition that is not suitable for the study drug
* 3. Known pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 7 days following injection
  Evaluation of Adverse Events (AE) Using CTCAE

SECONDARY OUTCOMES:
The diagnostic efficacy of 68Ga/64Cu-FAPI-XT injection in PET/CT imaging of patients with malignant solid tumor | 2 months following injection
  Accuracy (AC), sensitivity (SE), specificity (SP), positive predictive value (PPV)
Change in 'treatment strategy questionnaire' | 2 months following injection
  Referring physicians were asked to complete and return 2 questionnaires. The first assessed the existing treatment plan for the patient without the information from 68Ga/64Cu-FAPI-XT PET. The second inquired about intended management after receipt of the written clinical report and the 68Ga/64Cu-FAPI-XT PET images.

CONTACTS AND LOCATIONS:
Overall Officials: Ruimin Wang, Principal Investigator — the First Medical Center, Chinese PLA General Hospital
Locations (1):
- the First Medical Center, Chinese PLA General Hospital, Beijing, China